CLINICAL TRIAL: NCT04060277
Title: A Phase II Randomized, Placebo-Controlled, Multicenter Trial to Evaluate the Protective Function of CMV-MVA Triplex Vaccine in Adult Recipients of Haploidentical Hematopoietic Stem Cell Transplant
Brief Title: Triplex Vaccine in Preventing CMV Infection in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19065; NCI-2019-04888 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19065 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2019-07-29; First posted 2019-08-19 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid Cell Neoplasm; Hodgkin Lymphoma; Lymphoblastic Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Hematologic Neoplasms; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin | interventions — letermovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (letermovir, Triplex) (Experimental): Patients receive letermovir per SOC on days 7-100 and multi-peptide CMV-modified vaccinia Ankara vaccine IM on days 100 and 128 post-HCT.
  Interventions: Drug: Letermovir; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine
- Arm II (letermovir, placebo) (Active Comparator): Patients receive letermovir per SOC on days 7-100 and placebo IM on days 100 and 128 post-HCT.
  Interventions: Drug: Letermovir; Other: Placebo Administration

INTERVENTIONS:
Drug: Letermovir — Given as SOC
  Other Names: 2-((4S)-8-Fluoro-2-(4-(3-methoxyphenyl)piperazin-1-yl)-3-(2-methoxy-5-(trifluoromethyl)phenyl)-4H-quinazolin-4-yl)acetic Acid; AIC246; MK-8228; Prevymis
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine; Multi-antigen CMV-Modified Vaccinia Ankara Vaccine
  Arms: Arm I (letermovir, Triplex)
Other: Placebo Administration — Given IM
  Arms: Arm II (letermovir, placebo)

SUMMARY:
This phase II trial studies how well Triplex vaccine works in preventing cytomegalovirus (CMV) infection in patients undergoing a hematopoietic stem cell transplantation. CMV is a virus that may be carried for life and does not cause illness in most healthy individuals. However, in people whose immune systems are lowered (such as those undergoing stem cell transplantation), CMV can reproduce and cause disease and even death. The Triplex vaccine is made up of 3 small pieces of CMV deoxyribonucleic acid (DNA) (the chemical form of genes) placed into a weakened virus called modified vaccinia Ankara (MVA) that may help produce immunity (the ability to recognize and respond to an infection) and reduce the risk of developing complications related to CMV infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if CMV-MVA multi-peptide CMV-modified vaccinia Ankara vaccine (Triplex) reduces the frequency of clinically significant CMV reactivation in CMV positive (+) haploidentical hematopoietic cell transplantation (haploHCT) adult recipients from when letermovir (Prevymis) prophylaxis is stopped at day (d)100 until d180 post HCT.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of Triplex in vaccinated, haploHCT recipients by assessing the following: non-relapse mortality (NRM) at d180 post-HCT, severe (grade 3-4) acute graft versus host disease (GVHD), and grade 3-4 adverse events (AEs) (Common Terminology Criteria for Adverse Events [CTCAE] 5.0) probably or definitely related to the vaccination within 2 weeks from each vaccination at d180 post-HCT.

II. To characterize CMV related events in recipients of Triplex compared to placebo, by assessing time-to viremia (number of days from d100 to the date of >= 625 IU/mL), duration of viremia, recurrence of viremia, incidence of late CMV viremia/disease (>= 625 IU/mL, > 200 and =< 365 days post-HCT), use of antiviral drugs (triggered by clinically significant viremia), cumulative number of CMV specific antiviral treatment days.

III. To evaluate the impact of Triplex on transplant related outcomes up to d365 post-HCT by assessing the incidence of acute GVHD (aGVHD), chronic GVHD (cGVHD), relapse, non-relapse mortality, all-cause mortality, infections.

IV. To determine if Triplex increases levels, function and kinetics of CMV-specific T cell immunity in vaccinated compared to placebo treated, CMV seropositive HCT-recipients.

V. To determine whether vaccination induces adaptive natural killer (NK) cell population changes, and increase in the highly cytotoxic memory NKG2C+ NK cells.

VI. To compare GVHD biomarkers between the vaccine and placebo groups up to d365 post-HCT.

VII. To determine if immunity to 3 CMV antigens contained in the Triplex vaccine correlates with protection against CMV events, and if T-cell increases reflect vaccine response and exceed placebo immune response levels up to d365 post-HCT.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive letermovir per standard of care (SOC) on days 7-100 and multi-peptide CMV-modified vaccinia Ankara vaccine intramuscularly (IM) on days 100 and 128 post-HCT.

ARM II: Patients receive letermovir per SOC on days 7-100 and placebo IM on days 100 and 128 post-HCT.

After completion of study treatment, patients are followed up to 365 days post-HCT and then for an additional 2 years post-HCT.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* Planned peripheral blood stem cell (PBSC) or bone marrow (BM) HCT for the treatment of the following hematologic malignancies:

  * Lymphoma (Hodgkin and non-Hodgkin)
  * Myelodysplastic syndrome
  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status must be in hematologic remission by bone marrow and peripheral blood. Persistent lymphadenopathy on computed tomography [CT] or CT/positron emission tomography [PET] scan without progression is allowed.)
  * Acute myeloid leukemia in first or second remission
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase
  * Other hematologic malignancies judged appropriate by the clinical principal investigators (PIs), including chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis. Patients with multiple myeloma and those with non-malignant disease such as aplastic anemia are excluded

    * Adult cases of multiple myeloma (MM) are excluded as HCT is not standard of care for MM, and is only performed in very advanced cases with an associated high risk of relapse and NRM. Adults with aplastic anemia are excluded because their standard management includes T cell depletion with agents such as anti-thymocyte globulin (ATG), which is not permissible on this protocol. Patients undergoing a second haploHCT are not eligible (patients who have undergone a previous autologous HCT are eligible)
* Patients receiving myeloablative (MA) or reduced intensity conditioning (RIC) are allowed
* CMV seropositive (recipient)
* Planned related HCT with molecular 3/6 (haploidentical) intermediate/high resolution HLA donor allele matching
* Planned HCT with minimal to no-T cell depletion of graft
* Conditioning and immunosuppressive regimens according to institutional guidelines are permitted
* Negative serum or urine beta human chorionic gonadotropin (HCG) test (female patient of childbearing potential only) within two weeks of registration
* Seronegative for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and active hepatitis B virus (HBV) (surface antigen negative) within 2 months of registration and no history of disseminated cutaneous human papillomavirus (HPV) related disease
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for up to d90 post-HCT. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Any prior investigational CMV vaccine
* Experimental anti-CMV chemotherapy in the last 6 months
* Live attenuated vaccines (from the time of HCT to d70 post-HCT)
* Medically indicated subunit (Engerix-B for HBV; Gardasil for HPV) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections) (from the time of HCT to d70 post-HCT)
* Allergy treatment with antigen injections (from the time of HCT to d70 post-HCT)
* Alemtuzumab or any equivalent in vivo T-cell depleting agent (or CD34+ selection) (from the time of HCT to d70 post-HCT)
* Antiviral medications with known therapeutic effects on CMV such as ganciclovir (GCV)/valganciclovir (VAL), foscarnet (FOS), cidofovir, CMX-001, maribavir. Acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV) (from the time of HCT to d70 post-HCT)
* Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment EXCEPT Prevymis prophylaxis (prior to d100) (from the time of HCT to d70 post-HCT)
* Conditioning regimens d30 prior to trial participation and up to d180 post-HCT
* Disease-based radiation therapy (not total body irradiation) (from the time of HCT to d70 post-HCT)
* Other investigational product - concurrent enrollment in other clinical trials using any investigational new drugs (IND) with unknown effects on CMV or with unknown toxicity profiles is prohibited (from the time of HCT to d70 post-HCT)
* Other medications that might interfere with the evaluation of the investigational product (from the time of HCT to d70 post-HCT)
* Patients with active autoimmune conditions requiring systemic immunosuppressive therapy within the previous 5 years are not eligible
* Patients considered by PIs/protocol team to have a complicated prior therapy or HCT regimen, or who have a low survival probability (e.g., refractory leukemia and/or undergoing 2nd HCT)
* Poor risk disease/disease status including: chronic myeloid leukemia (CML) in blast crisis, acute myeloid leukemia (AML)/acute lymphoblastic leukemia (ALL) beyond 2nd remission, multiple myeloma, and aplastic anemia
* Pregnant women and women who are lactating. Triplex risks to pregnant women are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the administered vaccine, also breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., social/ psychological issues, etc.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2030-04-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the funding and development of a new successor multi-center trial, the study accrual was terminated early.
Period: Overall Study
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 48 [29 to 61] | 33 [24 to 59] | 48 [24 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cytomegalovirus (CMV) Events
Description: Cytomegalovirus (CMV) event was defined as CMV reactivation (DNAemia >625 IU/ml by qPCR), viremia treated by antivirals, or detection of CMV by tissue histology (end-organ disease), from Day 100 post-HCT to Day 180 post-HCT. Trial participants were quantitatively monitored for viremia, by plasma qPCR test once every two weeks (+/- 5d) from Day 100 to Day 180. CMV monitoring used standard qPCR clinical laboratory methods to evaluate CMV viral load and possible vaccine failure.
Time Frame: From Day 100 to Day 180 post-hematopoietic stem cell transplant (HCT)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Secondary Outcome: Non-Relapse Mortality at Day 180 Post-Transplant
Description: Non-relapse mortality (NRM) was defined as death without recurrent or progressive disease after transplant. NRM was estimated with the use of cumulative incidence curves, with relapse viewed as a competing risk.
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
percentage of participants | 0 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events

3. Secondary Outcome: Number of Participants With Severe (Grade 3-4) Acute Graft Versus Host Disease (GVHD) at Day 100
Description: Acute GVHD was assessed and graded according to the Keystone Consensus grading system (Przepiorka, D., et al., 1994 Consensus Conference on Acute GVHD Grading).
Time Frame: From time of transplant (Day 0) to Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

4. Secondary Outcome: Number of Grade 3-4 Adverse Events
Description: Adverse events probably or definitely related to the vaccination and modified vaccinia Ankara vector persistence were evaluated by NCI Common Terminology Criteria for Adverse Events v5.0.
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Number; unit: adverse events
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
adverse events | 0 | 0

5. Secondary Outcome: Duration of Viremia
Description: Duration of viremia was defined as the number of days from CMV qPCR >625 IU/mL to serum viral clearance (no detectable CMV DNA in serial blood samples).
Time Frame: From time of transplant (Day 0) to Day 200
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
days | NA [NA to NA] — lack of participants with events | NA [NA to NA] — lack of participants with events

6. Secondary Outcome: Number of Patients With Recurrence of CMV Viremia
Description: CMV viremia was defined CMV qPCR >625 IU/mL from samples collected within the past 7 days.
Time Frame: From time of transplant (Day 0) to Day 200
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

7. Secondary Outcome: Days From Transplant to ANC Engraftment
Description: Date of ANC engraftment was defined as the first date of ANC of ≥ 0.5 x 109/L achieved for 3 consecutive lab tests on 3 different days.
Time Frame: From time of transplant to date of ANC engraftment, up to Day 365.
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
days | 17 [14 to 18] | 16 [14 to 17]

8. Secondary Outcome: Cumulative Incidence of Acute GVHD
Description: Acute graft versus host disease is graded according to the 1994 Keystone Consensus Grading. The first day of acute GVHD onset was used to calculate the cumulative incidence. Relapse/death prior to onset was considered competing events.
Time Frame: From time of transplant (Day 0) to Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
percentage of participants | 25 [5 to 100] | 0 [NA to NA] — Insufficient number of participants with events

9. Secondary Outcome: Cumulative Incidence of Chronic GVHD at Day 365
Description: Cumulative incidence of Chronic GVHD (cGVHD) was estimated with the use of cumulative incidence curves. The first day of cGVHD onset was used to calculate the cumulative incidence. Relapse/death prior to onset was considered competing events.
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
percentage of participants | 33 [7 to 100] | 0 [NA to NA] — Insufficient number of participants with events

10. Secondary Outcome: Cumulative Incidence of Relapse at Day 365
Description: Cumulative incidence of relapse was estimated with the use of cumulative incidence curves, with death viewed as a competing risk.
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
percentage of participants | 0 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events

11. Secondary Outcome: Number Of Participants Died at Day 365
Description: Number of participants, who died due to all causes, at Day 365 post-transplant.
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

12. Secondary Outcome: Overall Survival at Day 365
Description: Estimates was calculated using the Kaplan-Meier method, Greenwood formula was used to calculate SE, and loglog transformation method was used to construct 95% confidence intervals. Each patient's vital status was monitored per clinical standard operating procedure. For this endpoint failure is defined as death (from any cause). Patients not experiencing a death event was censored at his/her date of last contact.
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
percentage of participants | 100 [100 to 100] | 100 [100 to 100]

13. Secondary Outcome: Non-Relapse Mortality (NRM) at Day 365
Description: as for outcome 2
Time Frame: From time of transplant (Day 0) to Day 365
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
percentage of participants | 0 [NA to NA] — Insufficient number of participants with events | 0 [NA to NA] — Insufficient number of participants with events

14. Secondary Outcome: Days From Transplant to Platelet Engraftment
Description: Date of platelet engraftment was defined as the first date of platelet value of ≥ 20 x 109/L achieved for 3 consecutive lab tests on 3 different days (without platelet transfusion in the previous 7 days).
Time Frame: From time of transplant to date of platelet engraftment, up to Day 365
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
Number analyzed (Participants) | 4 | 3
days | 23.5 [16 to 28] | 28 [18 to 33]

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were monitored/assessed at Day 100, 114, 128, 140, 180, 210-240, 270 and 365.
Arm/Group | Arm I (Letermovir, Triplex) | Arm II (Letermovir, Placebo)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Letermovir, Triplex) (N=4) | Arm II (Letermovir, Placebo) (N=3)
Fever (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Letermovir, Triplex) (N=4) | Arm II (Letermovir, Placebo) (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 2 (3)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 2 (3) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
motion sickness (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 1 (2)
White blood cell decreased (Investigations) | 3 (7) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (5) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT04060277/Prot_SAP_002.pdf
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT04060277/ICF_004.pdf